CLINICAL TRIAL: NCT07153484
Title: Assessment of Perception of Medical Professionals on Manikin-Based and Role-Play Simulation in Sudan 2025
Brief Title: Perception of Medical Professionals on Manikin-Based and Role-Play Simulation in Sudan
Status: Completed | Type: Observational
Sponsor: Research and Publication office (Other)
Responsible Party: Sponsor
Other Study IDs: 240012
Record Dates: First submitted 2025-09-02; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Simulation-based Medical Education
Keywords: Medical graduates and students; Role-playing simulation; Mannequin-based simulation; Simulation-based medical education; Sudan

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational Study

The goal of this observational study is to learn about the perceptions of Sudanese medical graduates and final-year students toward simulation-based medical education (SBME). The main question it aims to answer is:

Do medical professionals in Sudan view simulation-based training with mannequins and role-playing as helpful and effective?

Participants who had already experienced SBME completed an online survey about their learning experiences and confidence. A total of 408 responses were collected.

ELIGIBILITY:
Inclusion Criteria:

* Medical graduates (MBBS) and final-year medical students
* Previously underwent simulation-based training (during undergraduate education or professional development)

Exclusion Criteria:

* Graduates or students without exposure to simulation-based training
* Not located in Sudan during the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Medical graduates (MBBS) and final year medical students who previously underwent simulation based training, either during undergraduate education or their ongoing professional development.
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Participants' perceptions of simulation-based medical education | Jan 2025 - Apr 2025
  Participants' perceptions of simulation-based medical education (measured using the Student Satisfaction and Self-Confidence in Learning questionnaire, 5-point Likert scale).

CONTACTS AND LOCATIONS:
Overall Officials: Mona AA Hamad, Study Chair — Faculty of medicine and surgery National Ribat University, Khartoum,sudan; Azza Mustafa, Study Chair — National Ribat university; Ayman S Ahmed, Study Chair — National Ribat university; Emtithal AA Abdalrhman, Study Chair — Research and Publication Office, Karary University; Suhair Ali, Study Chair — Karary university,faculty of medicine; Eman Mohamed, Study Chair — Department of Hematology, Faculty of Medical Laboratory Sciences, International University of Africa.
Locations (1):
- Research and Publication Office, Khartoum, Khartoum State, Sudan

IPD SHARING:
Plan to Share IPD: No